CLINICAL TRIAL: NCT02132611
Title: Coronary Orbital Atherectomy System Study
Acronym: COAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-0005-P
Record Dates: First submitted 2014-05-06; First posted 2014-05-07 (Estimated); Results first posted 2016-10-27 (Estimated); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: CAD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diamondback 360® Coronary OAS Micro Crown (Experimental): Diamondback 360® Coronary Orbital Atherectomy System Micro Crown
  Interventions: Device: Diamondback 360® Coronary OAS Micro Crown

INTERVENTIONS:
Device: Diamondback 360® Coronary OAS Micro Crown — The Diamondback 360® Coronary OAS Micro Crown consists of a diamond-coated crown mounted to a shaft. The OAD ablates occlusive material in order to facilitate stent delivery. During orbit, forces press the crown against the coronary plaque, reducing calcified plaque on the vessel wall.

SUMMARY:
The purpose of the COAST clinical study data will be to utilize and to gain approval for commercializing the Micro Crown as part of the Coronary Orbital Atherectomy System (OAS).

DETAILED DESCRIPTION:
This is a prospective, single-arm, multi-center, global study designed to evaluate performance of the Diamondback 360® Coronary Orbital Atherectomy System Micro Crown (OAS Micro Crown) in treating de novo, severely calcified coronary lesions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 or older.
* Subjects must have a clinical indication for coronary intervention.
* CK and CK-MB must be less than or equal to the upper limit of lab normal value within 8 hours prior to the procedure.
* The target lesion must be a de novo coronary lesion that has not been previously treated with any interventional procedure.
* The target vessel must be a native coronary artery.
* The target vessel reference diameter must be >= 2.5mm and <= 4.0 mm.
* The lesion length must not exceed 40 mm.
* The target vessel must have a TIMI flow three (3) at baseline.
* The target lesion must have fluoroscopic, IVUS or OCT evidence of severe calcium deposit at the lesion site.
* The lesion must be crossable with the study guide wire.

Exclusion Criteria:

* Inability to understand the study requirements or has a history of non-compliance with medical advice.
* Unwilling to sign the COAST ICF.
* History of any cognitive or mental health status that would interfere with study participation.
* Currently enrolled in any other pre-approval investigational study.
* Female subjects who are pregnant or planning to become pregnant within the study period.
* Known hypersensitivity or contraindication to aspirin, heparin, ticlopidine or clopidogrel without adequate alternative medications.
* Known sensitivity to contrast media, which cannot be adequately pre-medicated.
* Diagnosed with chronic renal failure unless under hemodialysis, or has a serum creatinine level > 2.5 mg/dl.
* Experienced acute MI, STEMI or non-STEMI: CK-MB greater than the upper limit of lab normal value, within 30 days prior to index procedure.
* History of major cardiac intervention within 30 days.
* Evidence of heart failure
* History of a stroke or TIA within six (6) months.
* Active peptic ulcer or upper GI bleeding within six (6) months.
* History of bleeding diathesis or coagulopathy or intention to refuse blood transfusion, if one should become necessary.
* Concurrent medical condition with a life expectancy of < 12 months.
* History of immune deficiency.
* Uncontrolled insulin dependent diabetes.
* Evidence of active infections on the day of the index procedure.
* Subject has planned cardiovascular intervention within 60 days post index procedure.
* Subject is not an acceptable candidate for emergent CABG surgery.
* Subject with known allergy to atherectomy lubricant components such as soybean oil, egg yolk phospholipids, glycerin and sodium hydroxide.
* Subject with angiographically confirmed evidence of more than one (1) lesion requiring intervention, unless the treatment of the lesions is staged.
* Target lesion is located in a native vessel distal to anastomosis with a saphenous vein graft or LIMA/RIMA bypass.
* Target vessel has other lesions with greater than 50% diameter stenosis based on visual estimate or on-line QCA.
* Target vessel has angiographically visible or suspected thrombus.
* Target vessel has a stent from previous PCI.
* Target vessel appears to be or is excessively tortuous at baseline.
* Target lesion is an ostial location (within 5 mm of ostium) or an unprotected left main lesion.
* Target lesion is a bifurcation.
* Target lesion has a ≥ 1.5 mm side branch.
* Angiographic evidence of a dissection prior to initiation of OAD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg Stone, MD, Principal Investigator — Columbia University
Locations (17):
- United States (12):
  - Chandler Regional Medical Center and Mercy Gilbert Medical Center, Chandler, Arizona
  - North Florida Regional Medical Center, Gainesville, Florida
  - Palm Beach Gardens, Jupiter, Florida
  - Munroe Regional Health System, Inc., Ocala, Florida
  - Florida Hospital, Orlando, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Baptist Memorial Hospital/Stern Cardiovascular Foundation, Inc., Southaven, Mississippi
  - Mount Sinai Hospital New York, New York, New York
  - Columbia University Medical Center, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Duke University, Durham, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
- Japan (5):
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Saiseikai Yokohamashi Tobu Hospital, Yokohama, Kanagawa
  - Miyazaki Medical Association Hospital, Miyazaki, Miyazaki
  - Kyoto Katsura Hospital, Kyoto, Nishikyo-ku

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Redfors B, Sharma SK, Saito S, Kini AS, Lee AC, Moses JW, Ali ZA, Feldman RL, Bhatheja R, Stone GW. Novel Micro Crown Orbital Atherectomy for Severe Lesion Calcification: Coronary Orbital Atherectomy System Study (COAST). Circ Cardiovasc Interv. 2020 Aug;13(8):e008993. doi: 10.1161/CIRCINTERVENTIONS.120.008993. Epub 2020 Aug 6. PMID 32757661
- [Result] Martinsen BJ, Kumar K, Saito S, Sharma SK, Ikeno F, Fearnot NE, Shlofmitz RA, Thatcher R, Krucoff MW. Japan-USA Orbital Atherectomy for Calcific Coronary Lesions: COAST Study, Harmonization by Doing Proof-of-Concept. Cardiovasc Revasc Med. 2022 Apr;37:112-117. doi: 10.1016/j.carrev.2021.08.021. Epub 2021 Aug 26. PMID 34607786

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diamondback 360® Coronary OAS Micro Crown
Started | 100
Completed | 98
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Diamondback 360® Coronary OAS Micro Crown
Number analyzed (Participants) | 100
Age, Continuous [Mean (Full Range); unit: years] | 70.7 [45.1 to 89.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 71
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 2
  Black or African American | 2
  Japanese | 26
  Other | 2
  White | 65
  Unspecified | 3

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Cardiac Event (MACE)
Description: A Kaplan-Meier analysis was performed to determine the percent probability that a study participant is free from major adverse cardiac events at 30 days.
  30-Day MACE is composed of:
  * Cardiac death
  * Myocardial Infarction (MI) - defined as a Creatine Kinase Myocardial-Band Isoenzyme (CK-MB) level greater than three (3) times the Upper Limit of Lab Normal (ULN) value with or without new pathologic Q wave
  * Target Vessel Revascularization (TVR) - defined as a revascularization at the target vessel (inclusive of the target lesion) after the completion of the index procedure
Time Frame: 30 Days
Measure: Number (95% Confidence Interval); unit: Percent Probability of Freedom from MACE
Arm/Group | Diamondback 360® Coronary OAS Micro Crown
Number analyzed (Participants) | 100
Percent Probability of Freedom from MACE | 85.0 [78.0 to 92.0]

2. Secondary Outcome: Procedural Success
Description: Procedural success was defined as success in facilitating stent delivery with a residual stenosis of <50% and without the occurrence of an in-hospital MACE in de novo, severely calcified coronary lesions.
Time Frame: Participants were followed from baseline procedure through the duration of hospital stay, an average of 50.4 hours
Measure: Number (95% Confidence Interval); unit: percentage of procedures
Arm/Group | Diamondback 360® Coronary OAS Micro Crown
Number analyzed (Participants) | 100
percentage of procedures | 85.0 [76.5 to 91.4]

ADVERSE EVENTS:
Time Frame: 30 Days Post Procedure
Description: Serious Adverse Events reported by sites and adjudicated by the Clinical Events Committee.
Arm/Group | Diamondback 360® Coronary OAS Micro Crown
Serious Adverse Events (participants affected / at risk) | 27/100
Other Adverse Events (participants affected / at risk) | 9/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diamondback 360® Coronary OAS Micro Crown (N=100)
Acute MI, Q-wave (Cardiac disorders) | 2 (2)
Acute MI, non Q-wave (Cardiac disorders) | 12 (12)
Acute Congestive Heart Failure (Cardiac disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Coronary Artery Restenosis (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Carotid Artery Disease (Vascular disorders) | 1 (1)
Hematoma At Access Site, Not Requiring Intervention (Vascular disorders) | 1 (1)
Other Vascular Disorder (Vascular disorders) | 1 (1)
Gastrointestinal Bleeding (Gastrointestinal disorders) | 2 (2)
Renal Insufficiency (Renal and urinary disorders) | 1 (1)
Cardiac Death (Cardiac disorders) | 1 (1)
Non-Cardiac Death (General disorders) | 1 (1)
Abdominal Pain (General disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Chest Pain, Non-Cardiac (General disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Trauma (General disorders) | 1 (1)
Coronary Vessel Dissection Present (Surgical and medical procedures) | 7 (7)
Coronary Vessel Perforation Present (Surgical and medical procedures) | 2 (2)
Slow Flow or No Reflow Phenomena (Surgical and medical procedures) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diamondback 360® Coronary OAS Micro Crown (N=100)
Angiographic Complications (Surgical and medical procedures) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any previously unpublished information provided to the Investigators by the Sponsor is confidential and will remain the sole property of the Sponsor. The Investigator agrees to use this information only in accomplishing this study not use it for other purposes without the Sponsor's written consent. An Investigator can generate additional publication ideas based on the trial data. The Sponsor reserves the right to review the manuscript prior to submission in order to verify accuracy of the data.